CLINICAL TRIAL: NCT03107624
Title: Pre-infarction Angina and Culprit Plaque Characteristics in Patients With STEMI
Brief Title: Clinical Presentations Before AMI Onset and Coronary Atherosclerosis
Status: Completed | Type: Observational
Sponsor: Harbin Medical University (Other)
Responsible Party: Principal Investigator, Yu Bo, Director of Cardiology of The 2nd Affiliated Hospital of Harbin Medical University, Harbin Medical University
Other Study IDs: HMUOCT-PIA
Record Dates: First submitted 2017-03-22; First posted 2017-04-11 (Actual); Last update posted 2019-12-02 (Actual); Status verified 2018-05

CONDITIONS: Acute Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aimed to evaluate the incidence of preinfarction angina in AMI patients and test the hypothesis that different clinical presentations before AMI onset can affect coronary plaque morphologies in AMI patients .

DETAILED DESCRIPTION:
Patients with AMI who underwent primary percutaneous coronary intervention（PCI） and optical coherence tomography (OCT) examination is expected to be included in this study.Data about history were prospectively collected by a standard questionaire ,especially regarding the detail information about preinfarction angina.The basic clinical characteristics,angiographic and OCT findings are compared between patients with and without preinfarction angina.

ELIGIBILITY:
Inclusion Criteria：

1. Men or non-pregnant women >18 years of age and < 85 years of age;
2. Patients undergo cardiac catheterization for AMI;
3. Patients able to provide written informed consent.

Exclusion Criteria:

1. Patients cant afford medical history;
2. Cardiac shock；
3. Severe left ventricular dysfunction;
4. Left main disease;
5. Hepatic or kidney dysfunction;
6. OCT was performed after predilation;
7. Poor OCT image or massive thrombus.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: AMI patients
Sampling Method: Probability Sample
Enrollment: 305 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
Difference in culprit lesion morphologies assessed by OCT according to the presence or absence of PIA | baseline
  Plaque rupture was defined by the presence of a cavity formation in the plaque with a discontinuity of the fibrous cap. TCFA was defined as a lipid-rich plaque with a thin fibrous cap thickness of ≤ 65 um.Thrombus was identified by OCT as an irregular mass ≧0.25 mm in diameter protruding into the vessel lumen or attached to the surface of the vessel wall.Culprit lesion features in patients with PIA show a lower incidence of plaque rupture and TCFA compared to those without PIA.

SECONDARY OUTCOMES:
In-hospital outcomes after AMI. | baseline
  Infarct size was measured as the peak cardiac troponin I (cTnI) level.PIA is associated with lower infarct size and lower in-hospital mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Bo Yu, MD,PhD, Principal Investigator — The Second Affiliated Hospital of Harbin Medical University
Locations (1):
- The 2nd Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang, China

IPD SHARING:
Plan to Share IPD: No